CLINICAL TRIAL: NCT01692860
Title: Effects of Milk Protein Concentrate on Blood Pressure, Inflammation, Muscle Health During Weight Loss in Overweight/Obese Adults
Brief Title: Effects of Milk Protein Concentrate on Overall Health During Weight Loss in Overweight/Obese Adults
Acronym: S28
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph.D., Purdue University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1109011319
Record Dates: First submitted 2012-09-21; First posted 2012-09-25 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Sarcopenia; Metabolic Disease; High Blood Pressure
Keywords: the impact of a higher dairy-based protein diet in; combination with energy restriction on muscle health,; metabolic health (including blood pressure) in overweight; and obese, middle aged adults
MeSH Terms: conditions — Sarcopenia; Metabolic Diseases; Hypertension; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High protein consumption (Experimental): Intervention, energy restriction. This arm has a dietary protein intake of 1.5g/kg/d
  Interventions: Other: Energy Restriction
- Normal protein consumption (Placebo Comparator): Intervention, energy restriction. This arm has a dietary protein intake of .8g/kg/d
  Interventions: Other: Energy Restriction

INTERVENTIONS:
Other: Energy Restriction — Subjects consume 750 kcal/d of energy below their need

SUMMARY:
. The purpose of this study is to examine the effects of eating a larger amount of dairy-based protein on risk factors for metabolic syndrome

DETAILED DESCRIPTION:
Currently, over 47 million adults in the United States are known to have metabolic syndrome. Metabolic syndrome is comprised of a cluster of conditions including obesity, elevated cholesterol, high blood sugar, and high blood pressure. People with metabolic syndrome have an increased risk for the development of chronic diseases such as cardiovascular disease and diabetes. Recent studies have shown that a build-up of fat in the muscle of overweight and obese people may partially explain the link between metabolic syndrome and the development of chronic diseases. There is evidence to suggest that diets with a higher amount of protein can improve some aspects of metabolic syndrome, including the build-up of fat in muscle. The purpose of this study is to examine the effects of eating a larger amount of dairy-based protein on risk factors for metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

BMI: 25-38 ,male or female; age 35-65 y; weight stable (± 3 kg) during last 3 months; no acute illness; not diabetic, pregnant or lactating; not currently (or within last 3 months) following an exercise or weight loss program; non-smoking; not taking BP medication; not lactose intolerant,

Exclusion Criteria:

Subjects will be excluded if baseline protein intake is less than 0.6 or greater than 1.6 g•kg-1•d-1 Subjects will also be excluded if they have any chronic or acute condition which will increase risk of illness or injury during study participation as determined by our study physician such as high BP, high fasting glucose, metabolic syndrome, etc.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
weight loss | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph. D., Principal Investigator — Purdue University
Locations (1):
- Purdue University - Stone Hall 700 W State St, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Zhou J, Kim JE, Armstrong CL, Chen N, Campbell WW. Higher-protein diets improve indexes of sleep in energy-restricted overweight and obese adults: results from 2 randomized controlled trials. Am J Clin Nutr. 2016 Mar;103(3):766-74. doi: 10.3945/ajcn.115.124669. Epub 2016 Feb 10. PMID 26864362